# A Multi-center Cardiac PYP Scan Registry in Taiwan

#### NCT05593679

Date 2023-12-31

### **Objectives:**

This multi-center registry will collect the key cardiovascular data elements and set up PYP imaging database in Taiwan.

**Goal 1:** To standardize the imaging acquisition, analysis, interpretation and reporting.

**Goal 2:** To compare the clinical information and PYP imaging parameters in patients with suspected CA, to understand the real-world data in Taiwan.

### **Target Audience**

Every nuclear medicine department that performs PYP scan for cardiac amyloidosis

## **Project Design and Methods**

The investigators will retrospectively and prospectively collect total 1,000 PYP scans that had been performed on suspected or diagnosed ATTR-CM patients in Taiwan and follow-up at least 1 year. All patients are enrolled based on clinical suspicions such as "red-flag" signs using ultrasound, NT-pro BNP and clinical data according to the diagnostic algorithms. Due to the diverse consensus or guidelines' recommendations, some physicians may arrange PYP scans before AL exclusion. In patients with Grade 2 and 3 PYP myocardial uptake, genetic testing is arranged, serum and urine AL tests results should be confirmed. All the clinical information including demographic data, lab, echocardiography, or other cardiac imaging (ex. MRI) will be collected. The clinical information, genetic testing and imaging parameters derived from PYP scans (visual scores, and H/CL ratios) will be analyzed and compared by t-test or ANOVA based on clinical diagnosis and PYP grades.